CLINICAL TRIAL: NCT04757532
Title: Study of Exposure to Substances Prohibited by the World Anti-Doping Agency in Healthy Volunteers.
Acronym: ESPAMA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IMIMFTCL/ESPAMA
Record Dates: First submitted 2021-02-14; First posted 2021-02-17 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-02

CONDITIONS: Healthy Volunteers
Keywords: Anti-doping control; Bupropion; Anastrozole; Danazol; Chlorthalidone; Testosterone
MeSH Terms: interventions — Bupropion; Anastrozole; Testosterone Propionate; Danazol; Chlorthalidone

STUDY DESIGN:
Intervention Model Description: Single-center, non-randomized, unblinded, uncontrolled clinical trial in healthy male volunteers, at a single dose of the five study drugs (bupropion, anastrozole, testosterone cyclopentylpropionate, danazol and chlorthalidone).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Bupropion (Experimental): Subjects receive a single-dose treatment. Urine samples will be collected until 3 days after administration in 6 fractions: 0-4h, 4-8h, 8-12h, 12-24h, 24-48h, 48-72h post-administration.
  Interventions: Drug: Bupropion
- Anastrozole (Experimental): Subjects receive a single-dose treatment. Urine samples will be collected until 7 days after administration in 7 fractions: 0-24h, 24-48h, 48-72h, 72-96h, 96-120h, 120-144h, 144-168h post-administration.
  Interventions: Drug: Anastrozole
- Testosterone cyclopentylpropionate (Experimental): Subjects receive a single-dose treatment. Urine samples will be collected until 20 days after administration in 20 fractions: first urine of the day, every day.
  Interventions: Drug: Testosterone cyclopentylpropionate
- Danazol (Experimental): Subjects receive a single-dose treatment. Urine samples will be collected until 2 days after administration in 6 fractions: 0-4h, 4-8h, 8-12h, 12-24h, 24-36h, 36-48h post-administration.
  Interventions: Drug: Danazol
- Chlorthalidone (Experimental): Subjects receive a single-dose treatment. Urine samples will be collected until 3 days after administration in 4 fractions: 0-12h, 12-24h, 24-48h y 48-72h post-administration.
  Interventions: Drug: Chlorthalidone

INTERVENTIONS:
Drug: Bupropion — 300 mg of bupropion hydrochloride (1 tablet) administered orally in a single dose.
  Other Names: Elontril®
  Arms: Bupropion
Drug: Anastrozole — 1 mg of anastrozole (1 tablet) administered orally in a single dose.
  Other Names: Anastrozol Mylan®
  Arms: Anastrozole
Drug: Testosterone cyclopentylpropionate — 100 mg of testosterone cyclopentylpropionate (equivalent to 70 mg of testosterone) administered via intramuscular injection in a single dose (2 mL).
  Other Names: Testex prolongatum®
  Arms: Testosterone cyclopentylpropionate
Drug: Danazol — 200 mg of danazol (1 capsule) administered orally in a single dose.
  Other Names: Danatrol®
  Arms: Danazol
Drug: Chlorthalidone — 50 mg of chlorthalidone (1 tablet) administered orally in a single dose.
  Other Names: Higrotona®
  Arms: Chlorthalidone

SUMMARY:
Background:

The use of stimulants such as bupropion, enzyme inhibitors such as anastrozole, androgens such as testosterone, antigonadotropins such as danazol, and diuretics such as chlorthalidone have been reported in urine drug testing programs for a wide variety of applications, including anti-doping tests in sport. These substances are subject to screening studies by the World Anti-Doping Agency (WADA). Anastrozole, chlorthalidone, testosterone and danazol are included on the WADA list of prohibited substances, while bupropion is included in the 2020 follow-up schedule of substances.

This study aims to characterize the urinary excretion patterns of these substances following the administration of a single dose of each drug at a recommended therapeutic dose.

Hypothesis:

The administration of bupropion, anastrozole, testosterone, danazol or chlorthalidone in healthy subjects allows the generation of detectable concentrations of the drug in urine using the liquid chromatography technique coupled to mass spectrometry (LC-MS). Positive urine samples will enable to identify analytical strategies for doping control.

Objectives:

Primary objective: To measure the concentrations of various drugs (anastrozole, bupropion, chlorthalidone, danazol and testosterone) and their metabolites in urine for anti-doping control samples. The detection of new metabolites excreted in urine for longer periods of time than conventional metabolites will improve the ability to detect the abuse of anabolic steroids in sport.

Secondary objective: To assess safety and tolerability of the drugs used.

Methods:

Phase I, unicentric, open, non-randomized, non-controlled clinical trial, with 5 parallel treatment conditions (anastrozole, bupropion, chlorthalidone, danazol and testosterone) administered in a single dose to male healthy volunteers (total n=11).

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers aged between 18 and 50 years.
* Able to understand and accept the trial procedures and able to sign an informed consent.
* History and physical examination that demonstrate not presenting organic or psychiatric disorders.
* ECG, blood and urine tests performed before the experimental session within normal limits. Minor or occasional variations of these limits will be allowed if, in the opinion of the Principal Investigator and taking into account the state of science, they have no clinical significance, do not pose a risk to the subject and do not interfere in the product evaluation. These variations and their non-relevance will be specifically justified in writing.
* Body mass index (weight/height^2) between 19 and 27 kg/m2 and weight between 50 and 100 kg. BMI of 27-28 kg/m2 may be included according to Principal Investigator's criteria.

Exclusion Criteria:

* Failure to meet inclusion criteria.
* History of allergy, idiosyncrasy, hypersensitivity or adverse reactions to the active substance or any of the excipients. Lactose intolerance. Serious adverse reactions to any drug.
* Contraindications to treatment with study drugs (according to the respective summary of product characteristics, SmPC). Especially history or presence of breast cancer, liver cancer, and suspected or confirmed prostate carcinoma.
* History or current presence of prostate syndrome symptoms: frequent urination (both day and night), difficulty in starting urination, weak or discontinuous urinary stream, feeling of incomplete bladder emptying, or benign prostatic hyperplasia diagnosis.
* Levels of prostate specific antigen (PSA) out of normal range for subject's age, in those receiving anastrozole, testosterone or danazol.
* Clinical background or evidence of gastrointestinal, hepatic, renal disorder or others that may involve an alteration of the absorption, distribution, metabolism or excretion of the drug.
* Clinical background or evidence of psychiatric disorders, alcoholism, drug abuse or habitual consumption of psychoactive drugs.
* Having participated in another clinical trial with medication in the three months prior to the start of the study.
* Having suffered some organic disease or major surgery in the six months prior to the start of the study.
* Clinical background or evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological, neurological, dermatological or other acute or chronic diseases that, in the opinion of the Principal Investigator or the collaborators designated by him/her, may pose a risk to the subjects or may interfere with the objectives of the study. Especially history of venous thrombosis or thromboembolic disorders, thrombophilic alteration, edema, hypercalcemia, polycythemia, nephrosis, liver disease with altered liver function tests and porphyria.
* Having taken medication regularly in the month prior to the study sessions, including vitamins, herbal remedies or dietary supplements. Treatment with a single dose of symptomatic medication in the week prior to the study sessions will not be a reason for exclusion if it is assumed that the drug has been completely eliminated on the day of the experimental session.
* Smokers of more than 20 cigarettes a day in the 3 months before the study.
* Consumption of more than 40 g of alcohol daily.
* Consumers of more than 5 coffees, teas, cola drinks, or other stimulant drinks or with xanthines daily in the 3 months prior to the study start.
* Being unable to understand the nature, consequences of the trial and the procedures that are asked to follow.
* Positive serology for hepatitis B, C or HIV.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Urine concentration of bupropion metabolites | 0-4 h (hours), 4-8h, 8-12h, 12-24h, 24-48h and 48-72h post-administration
  Concentration of bupropion metabolites in each fraction of urine samples
Urine concentration of anastrozole metabolites | 0-24 h (hours), 24-48h, 48-72h, 72-96h, 96-120h, 120-144h and 144-168h post-administration
  Concentration of anastrozole metabolites in each fraction of urine samples
Urine concentration of testosterone metabolites | 0-20 days post-administration (24-hour fractions)
  Concentration of testosterone metabolites in each fraction of urine samples
Urine concentration of danazol metabolites | 0-4 h (hours), 4-8h, 8-12h, 12-24h, 24-36h and 36-48h post-administration
  Concentration of danazol metabolites in each fraction of urine samples
Urine concentration of chlorthalidone metabolites | 0-12 h (hours), 12-24h, 24-48h and 48-72h post-administration
  Concentration of chlorthalidone metabolites in each fraction of urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Aldea Perona, MD PhD, Principal Investigator — IMIM (Hospital del Mar Medical Research Institute)
Locations (1):
- IMIM (Hospital del Mar Medical Research Institute), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No